CLINICAL TRIAL: NCT03285269
Title: Extension of the Rapid Ultrasound for Shock and Hypotension to Evaluate Volume Responsiveness
Brief Title: Extension of the RUSH Protocol for Volume Responsiveness
Status: Withdrawn | Type: Observational
Why Stopped: Study was not initiated because it was not approved by KPSC IRB.
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: ERUSH-001
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Shock
Keywords: shock; ultrasound
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Shock Group: Patients presenting with signs and symptoms of shock will undergo the E-RUSH ultrasound protocol and bioreactance before and after a passive leg raise maneuver.
  Interventions: Diagnostic Test: Ultrasound Protocol; Device: Bioreactance; Procedure: Passive Leg Raise

INTERVENTIONS:
Diagnostic Test: Ultrasound Protocol — Ultrasound of the inferior vena cava, heart and lungs.
Device: Bioreactance — Bioreactance assessment using Cheetah Bioreactance Device (FDA Approved). Bioreactance is a non-invasive measure of cardiac output.
Procedure: Passive Leg Raise — A passive leg raise involves placing the patient supine and raising the legs to simulate an intravenous fluid bolus.

SUMMARY:
The current study plants to create a patient registry of patients who present to the emergency department with signs and symptoms of shock and evaluate the ability of a multi-step cardiopulmonary ultrasound protocol to determine the need for fluid therapy.

DETAILED DESCRIPTION:
Background & Motivation: Non-traumatic shock accounts for millions of emergency department visits every year and is a significant burden on the health care system making rapid identification and treatment essential. For decades the Rapid Ultrasound in Shock and Hypotension (RUSH) exam has been employed to help determine the etiology of non-traumatic shock in the ED setting. The RUSH exam does not answer other critical questions such as the need for additional fluid resuscitation. The current study hypothesizes that by include a step-wise cardiopulmonary algorithm the RUSH exam can be extended (E-RUSH) to accurately determine the need for additional fluid therapy.

Study Design: Prospective Observational Study in two urban Emergency Departments with a combined annual census of >111,000.

Population: ED patients exhibiting signs of shock definied by a systolic blood pressure < 100 mmhg, MAP < 65, persistent tachycardia, mottled skin, or lactate >2mmol either at presentation or during ED stay will be included. Exclusion criteria will be inability to consent, external factors preventing ultrasound examination, age less than 18, pregnancy, incarceration, arrhythmia, cardiac arrest, or treating physician gestalt that the patient is not in shock.

Protocol: The E-RUSH protocol will include ultrasound exams of the IVC, heart and lungs as described in the RUSH protocol but will also evaluate cardiac output, IVC collapsibility, and presense of B-lines on lung ultrasound. At the time of ultrasound measuresments a bioreactance device will be applied. Bioreactance measurements and ultrasound measurement of cardiac output will be recorded pre and post a passive straight leg raise test. All charts will be reviewed by two experts who are blinded to ultrasound and bioractance measurements. When possible the protocol will be repeated 1-2 hours later or after initial interventions in order to provide trend data.

Data Analysis: Volume responsivness as assessed by the E-RUSH will be defined a priori using a step-wise flow diagram that combines IVC, lung and cardiac ejection fraction and output measurements (see research plan for details). Determination of volume responsiveness by the bioreactance device will be defined by manufacturer protocal. Determination of volume responsiveness by expert review will be by a standard abstraction form with agreement of both expert reviewers. Descriptive statistics will be performed to determine the test characteristics of the ultrasound protocol to predict volume responsiveness. Given the lack of a universally agreed upon gold standard for volume responsiveness, we will determine test characteristics for E-RUSH using the bioreactance device as a reference standard and using expert review as a second reference standard separately.

FACILITY RESOURCES The study facilities are in San Diego California, with a combined emergency department census of over 111,000 patients per year. The emergency departments of the facilities are equipped with portable bedside ultrasound machines, CT and MRI, 24 hour laboratory testing and an integrated electronic medical record system. Emergency medicine and family medicine residents rotate through both emergency departments. Both departments are stroke receiving centers and level 3 trauma centers.

Research Databases An important aspect of the KPSC managed care environment is its integrated approach to the delivery of medical care. This approach depends on, and therefore facilitates, the development and maintenance of a large number of databases, linkable through a unique identification key. These databases include those that track membership, encounters, laboratory, claims, pharmaceutical dispensations and others. The address information is annually geo-coded to the census block level, providing linkage to census-based group-level information about socio-economic status.

Each of the KPSC clinical operations systems are updated in real-time, facilitating our ability to create near real-time research databases. Our Membership database captures demographic (e.g., name, date of birth, gender, race/ethnicity, etc.) and benefit information for over 12 million active and former members, and is updated on a weekly basis. The utilization database captures outpatient and hospital encounters (e.g., diagnoses, procedures, etc.), member claims submitted from outside hospitals (usually with up to 3-month delay), and care provided at home, skilled nursing and hospice facilities. This database is updated weekly. Outpatient and inpatient pharmacy databases track medication orders and dispenses, and are updated either daily or monthly depending on the source system. Death information is derived from multiple sources including KP hospital and membership data, as well as two external sources from California State and Social Security Administration death files. The state death records lag about one to two years for date and underlying cause of death and between two and three years for all causes listed on the death certificate.

SCIENTIFIC ENVIRONMENT Biostatistical expertise is provided by a Biostatistics Unit that consists of statisticians, programmers, natural language specialists, database developers and administrators. The Unit provides services including statistical consultation, data analysis, data extraction, disease identification based on free-texts and data management for research projects. In addition, the Unit is responsible for creating many of the research data bases used. All Unit employees have SAS programming skills and years of experience in conducting broad and varied research. The Biostatistics Unit supports more than 300 research projects annually.

Oversight of Research at KPSC KPSC has an Institutional Review Board (IRB) under the Medical Director of Operations for the Southern California Permanente Medical Group. The IRB is charged with the protection of human subjects through the oversight of all investigators and their research projects in Kaiser Permanente Southern California. Compliance with the minimum Federal standards for the protection of human subjects in research is demonstrated by a Federal Wide Assurance (FWA) held through the Kaiser Foundation Research Institute. The IRB also acts as the KPSC HIPAA privacy board.

Ethics Kaiser Permanente - Southern California (KPSC) shall obtain written evidence of review and approval from our independent ethics committee (IRB) of the protocol, informed consent forms, evidence of partial waiver, and all other documents requiring IRB review and approval prior to the initiation of the project.

1. RISKS TO THE SUBJECTS

   1. Human Subjects Involvement and Characteristics Describe the proposed involvement of human subjects in the work outlined in the Research Design and Methods section.

      The study population are ED patients exhibiting signs of shock definied by a systolic blood pressure < 100 mmhg, MAP < 65, persistent tachycardia, mottled skin, or lactate >2mmol either at presentation or during ED stay will be included. Exclusion criteria will be inability to consent, external factors preventing ultrasound examination, age less than 18, pregnancy, incarceration, traumatic mechanism, arrhythmia, cardiac arrest, or treating physician gestalt that the patient is not in shock. Our goal is to enroll a total of 50 patients.

      This study will not recruit subjects defined as vulnerable populations. Individuals age less than 18 and pregnant women will be excluded as noted in the exclusion criteria.
   2. Sources of Materials

   The following data will be obtained from the patient:
   * Consent Form
   * ultrasound will be used to perform visual assessment of the patient's inferior vena cava
   * Variables including but not limited to: systolic blood pressure, MAP, persistent tachycardia, mottled skin, or lactate status, age, pregnancy status, arrhythmia, cardiac arrest,
   * "Electronic Health Data" - All charts will be reviewed by two experts who are blinded to ultrasound and bioractance measurements.
   * Bioreactance measurements and ultrasound measurement of cardiac output will be recorded pre and post a passive straight leg raise test.

   The data collected will be linked/coded using a study identification number (SID) and only KPSC study team members and persons directly involved in recruitment will have access to the key that identifies individual subjects.
2. ADEQUACY OF PROTECTION AGAINST RISKS

   1. Recruitment and Informed Consent We will obtain a waiver to access and use the EHR data for case/patient identification. The waiver will be used to identify patients in order approach patients regarding the study and to obtain consent. Study personnel will screen the ED tracking board and communicate with ED providers to find patients meeting inclusion criteria. Upon identification study personnel, will approach patient in the private exam room to obtain informed consent in person.

      The study will not recruit anyone less than 18 or women who are pregnant. However, due to the rich diversity of Kaiser Permanente's membership in Southern California, Spanish speakers will be recruited. All materials and forms will be translated to Spanish to include all Spanish speaking/reading potential participants. Consent forms will be stored securely onsite and a study database will be maintained. All patients will be provided a copy of the consent form.
   2. Protection Against Risk Names and other identifying information on participants will be obtained for record keeping purposes only and no participants will be identified in any forms or reports from this study. Survey and clinical data will only be shared internally among KPSC study team members and only persons directly involved in recruitment will have access to the key that identifies individual subjects. Transfer of data if needed will be via encrypted email.
3. POTENTIAL BENEFITS OF THE PROPOSED RESEARCH TO THE SUBJECTS AND OTHERS The immediate benefit to the participant is none. However, If the E-RUSH protocol proves accurate and useful, it has the potential to improve patient care and safety and a vulnerable and high risk population. There are no high-risk aspects of the proposed work.
4. IMPORTANCE OF THE KNOWLEDGE TO BE GAINED There are no high-risk aspects of the proposed work. The importance of the current study presents an innovative algorithm that my further demonstrate the ability of ultrasound to be useful in the shock patient to determine fluid needs. If an algorithmic approach using bedside ultrasound proves accurate in titrating fluid resuscitation, it could reduce complications of under resuscitation (organ failure) and over resuscitation (pulmonary edema, third spacing and abdominal compartment syndrome). Avoidance of complications would have downstream benefits such as reduced length of stay, reduced mortality, and reduced burden on the healthcare system.
5. DATA AND SAFETY MONITORING PLAN Our study will not be a clinical trial. All the information and/or databases will be password protected to ensure security of the PHI contained in the data systems. Study data access that would identify participants will be tightly controlled and limited to authorized individuals using the follow safeguards: roles and privileges, defined data owners, automatic log off and lockouts, field level hide, read only, or read-write permission at user level, encryption of data transfers, and limited/controlled delete capabilities. Standard backup procedures will be employed at Kaiser Permanente, where data will be backed up nightly to a secured disk based storage system and then offloaded to a robotic tape library system, with tapes rotated offsite for additional level of protection. This ensures against data loss in the event of a local systems failure or natural disaster.

ELIGIBILITY:
Inclusion Criteria:

* ED patients exhibiting signs of shock definied by a systolic blood pressure < 100 mmhg, MAP < 65, persistent tachycardia, mottled skin, or lactate >2mmol either at presentation or during ED stay will be included

Exclusion Criteria:

* Exclusion criteria will be inability to consent, external factors preventing ultrasound examination, age less than 18, pregnancy, incarceration, arrhythmia, cardiac arrest, or treating physician gestalt that the patient is not in shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the one of two urban emergency department with signs and symptoms of shock.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Test Characteristics of the E-RUSH Protocol to Predict Fluid Responsiveness | 1 year
  Will determine sensitivity and specificity of a step-wise cardiopulmonary approach to determine fluid responsivness.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Fields, MD, Principal Investigator — Kaiser Permanenete

IPD SHARING:
Plan to Share IPD: No
Not planning to share IPD

REFERENCES:
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Bentzer P, Griesdale DE, Boyd J, MacLean K, Sirounis D, Ayas NT. Will This Hemodynamically Unstable Patient Respond to a Bolus of Intravenous Fluids? JAMA. 2016 Sep 27;316(12):1298-309. doi: 10.1001/jama.2016.12310. PMID 27673307
- [Background] Boyd JH, Forbes J, Nakada TA, Walley KR, Russell JA. Fluid resuscitation in septic shock: a positive fluid balance and elevated central venous pressure are associated with increased mortality. Crit Care Med. 2011 Feb;39(2):259-65. doi: 10.1097/CCM.0b013e3181feeb15. PMID 20975548
- [Background] Corl KA, George NR, Romanoff J, Levinson AT, Chheng DB, Merchant RC, Levy MM, Napoli AM. Inferior vena cava collapsibility detects fluid responsiveness among spontaneously breathing critically-ill patients. J Crit Care. 2017 Oct;41:130-137. doi: 10.1016/j.jcrc.2017.05.008. Epub 2017 May 12. PMID 28525778
- [Background] Monnet X, Marik PE, Teboul JL. Prediction of fluid responsiveness: an update. Ann Intensive Care. 2016 Dec;6(1):111. doi: 10.1186/s13613-016-0216-7. Epub 2016 Nov 17. PMID 27858374
- [Background] Oord M, Olgers TJ, Doff-Holman M, Harms MP, Ligtenberg JJ, Ter Maaten JC. Ultrasound and NICOM in the assessment of fluid responsiveness in patients with mild sepsis in the emergency department: a pilot study. BMJ Open. 2017 Jan 27;7(1):e013465. doi: 10.1136/bmjopen-2016-013465. PMID 28132006
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169